CLINICAL TRIAL: NCT00229021
Title: A Multicenter, Double-Blind, Randomized, Phase 3 Study of Doripenem Verus a Comparator Antibiotic in the Treatment of Complicated Lower Urinary Tract Infection or Pyelonephritis
Brief Title: Doripenem in the Treatment of Complicated Lower Urinary Tract Infection or Pyelonephritis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Collaborators: Peninsula Pharmaceuticals, Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR005404
Record Dates: First submitted 2005-09-27; First posted 2005-09-29 (Estimated); Last update posted 2011-06-10 (Estimated); Status verified 2010-04

CONDITIONS: Urinary Tract Infections; Pyelonephritis
Keywords: Complicated Urinary Tract Infection; Pyelonephritis
MeSH Terms: conditions — Urinary Tract Infections; Pyelonephritis

INTERVENTIONS:
Drug: doripenum

SUMMARY:
The purpose of this study is to compare the microbiological cure rate of doripenem versus a comparator antibiotic in the treatment of patients with complicated urinary tract infection or pyelonephritis. The study will also characterize the safety and tolerability of treatment with doripenem in patients with complicated urinary tract infection or pyelonephritis.

DETAILED DESCRIPTION:
Doripenem is an antibiotic medication not yet approved by the US FDA. This is a phase 3, multi-center, randomized, prospective, double-blind study of doripenem versus comparator in the treatment of complicated lower urinary tract infections (UTI) or pyelonephritis in adults. After the screening, patients are randomized to receive either doripenem or comparator. Patients are hospitalized, but subsequently, patients may be treated as outpatient or through home-based therapy at the investigators' discretion. Conventional laboratory data are collected from all patients at specified times throughout the study. The primary endpoint is microbiological response measured at test of cure visit. The patients receive either doripenum or comparator; duration of therapy is 10 days.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of complicated lower urinary tract infection or pyelonephritis

Exclusion Criteria:

* Women who are pregnant, nursing or of child-bearing potential and not using a medically accepted, effective method of birth control
* History of moderate or severe hypersensitivity reactions to antibiotic medications

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 741 (Actual)
Dates: Start 2003-12; Study Completion 2006-03 (Actual)

PRIMARY OUTCOMES:
Microbiological response measured at test of cure visit at early follow-up.

SECONDARY OUTCOMES:
Clinical response (cure) assessed at early follow-up visit. Proportion of patients with sustained microbiological and clinical response measured at late follow-up visit. Safety evaluations will be conducted throughout the study.

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development, L.L. C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.

REFERENCES:
- [Derived] Redman R, Damiao R, Kotey P, Kaniga K, Davies T, Naber KG. Safety and efficacy of intravenous doripenem for the treatment of complicated urinary tract infections and pyelonephritis. J Chemother. 2010 Dec;22(6):384-91. doi: 10.1179/joc.2010.22.6.384. PMID 21303745
- [Derived] Kaniga K, Flamm R, Tong SY, Lee M, Friedland I, Redman R. Worldwide experience with the use of doripenem against extended-spectrum-beta-lactamase-producing and ciprofloxacin-resistant Enterobacteriaceae: analysis of six phase 3 clinical studies. Antimicrob Agents Chemother. 2010 May;54(5):2119-24. doi: 10.1128/AAC.01450-09. Epub 2010 Mar 8. PMID 20211892
- [Derived] Zhanel GG, Ketter N, Rubinstein E, Friedland I, Redman R. Overview of seizure-inducing potential of doripenem. Drug Saf. 2009;32(9):709-16. doi: 10.2165/00002018-200932090-00001. PMID 19670912
- See also: A Multicenter, Double-blind, Randomized, Phase 3 Study to Compare the Safety and Efficacy of Intravenous Doripenem and Levofloxacin in Complicated Lower Urinary Tract Infection or Pyelonephritis — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=642&filename=CR005404_CSR.pdf